CLINICAL TRIAL: NCT06442813
Title: Effects Of Emotional Freedom Technique and Hypermesis Gravidarum
Acronym: PREGNANCY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Merve Meşedüzü, LECTURER, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-54022451-050.05.04-91178; MMeseduzu (Other: BezmialemVU)
Record Dates: First submitted 2024-01-12; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Hyperemesis Gravidarum; Pregnancy
Keywords: hyperemesis gravidarum; quality life; pregnancy; Emotional Freedom Techniques
MeSH Terms: conditions — Hyperemesis Gravidarum

STUDY DESIGN:
Intervention Model Description: EXPERIMENTAL GROUP First Stage: Determining the groups by randomization method and filling out the data collection forms for the groups (pre-test).
  Second Stage: Training pregnant women in the control group on the management of standard hyperemesis gravidarum (training content will be prepared and opinions will be obtained from 3 experts in the field).
  For the intervention group, pregnant women were given a session with EFT (Average: 40-60 minutes) and a program was created for the pregnant woman to do affirmations in between depending on her condition (Positiveness with EFT strokes 3 times a day).
  Third Stage: After 15 days, it is planned to conduct post-tests for both groups and
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERİMENTAL GROUP (Experimental): First Stage: Determining the groups by randomization method and filling out the data collection forms for the groups (pre-test).
  Second Stage: Training pregnant women in the control group on the management of standard hyperemesis gravidarum (training content will be prepared and opinions will be obtained from 3 experts in the field).
  For the intervention group, pregnant women were given a session with EFT (Average: 40-60 minutes) and a program was created for the pregnant woman to do affirmations in between depending on her condition (Positiveness with EFT strokes 3 times a day).
  Third Stage: After 15 days, it is planned to conduct post-tests for both groups and complete the study. In the final stage, pregnant women's questions will be answered, counseling will continue where deemed necessary, and prepared training booklets will be given to pregnant women
  Interventions: Behavioral: EFT GROUP
- CONTROL GROUP (No Intervention): Pregnant women diagnosed with hyperemesis gravidarum (HG) who meet the inclusion criteria for the study will constitute the control group. Providing training to the control group only for HG management (training content will be prepared and opinions will be obtained from 3 experts in the field).

INTERVENTIONS:
Behavioral: EFT GROUP — One times one pregnancy
  Other Names: emotıonal free technıcal
  Arms: EXPERİMENTAL GROUP

SUMMARY:
The purpose of this clinical study is to determine whether EFT (Emotional Freedom Techniques) is effective in alleviating nausea and vomiting in pregnant women with hyperemesis. Additionally, the study aims to gather information on the safety of EFT application. The primary questions it seeks to answer are:

Does EFT reduce nausea and vomiting in pregnant women with hyperemesis? Is EFT applicable for use in pregnant women with hyperemesis? Researchers will compare the effectiveness of EFT to traditional nursing education on non-pharmacological interventions for preventing nausea and vomiting in pregnant women with hyperemesis.

Participants:

Pre-EFT application survey scale questions will be asked to the pregnant women with hyperemesis.

EFT will be applied once by the researcher to the pregnant women with hyperemesis.

For control, the same survey scale questions will be asked to the same pregnant women two days after the EFT application for post-test purposes.

For control, the same survey scale questions will be asked to the same pregnant women seven days after the EFT application for post-test purposes.

The same procedures will be applied in the same manner to the control group that will receive education.

DETAILED DESCRIPTION:
Type of Research: It is planned to be randomized, controlled and experimental. Place and Characteristics of the Research: The research will be carried out in the women health and diseases service and Gynecology polyclinics of Bezmialem Vakif University Faculty of Medicine Central Hospital.

Population and Sample of the Research:The sample size was determined as a minimum of 74 people in total using the G Power 3.1 method. The effect size was determined using the t test values in the reference study in which the scale was used with a similar patient group.

Criteria for Inclusion in the Study:Pregnant women who are between 6 and 14 weeks of gestation, aged between 20 and 40 years old, and have complaints of nausea and vomiting are eligible for the study. These participants should report their discomfort as 5 or above on the VAS scale. Additionally, they must not have been diagnosed with a high-risk pregnancy or any psychological disorders. Lastly, they must voluntarily agree to participate in the study.

Criteria for Exclusion from the Study: Exclusion criteria are the presence of coordination and language problems in the pregnant woman and her desire to leave the study at any time or not to participate.

Survey Scales Descriptive Information Form: The pregnancy information form, prepared in line with the literature review conducted by the researchers, includes socio-demographic (age of the pregnant woman, education and employment status, income level, family type and place of residence), obstetric (current gestational week and pregnancy history), psychosocial information. It consists of questions about social and medical history (pregnancy desire), whether there is a chronic disease) and VAS Scale. VAS is a measurement tool used to measure both pain intensity and pain relief, which is simple, effective and repeatable and requires minimal tools.

2. Pregnancy-Specific Nausea and Vomiting Severity Scale (PUQE-24): its form specific to the pregnancy period that evaluates nausea and vomiting for the last 12 hours. It was later reported that it would be more appropriate to evaluate the last 24 hours for clinical use, as the last 12 hours sometimes include the sleep period in terms of nausea and vomiting in pregnant women. Thereupon, the Pregnancy-Unique Quantification of Emesis (PUQE-24) Scale was developed and evaluate the severity of pregnancy-specific nausea and vomiting in the last 24 hours. Its Turkish validity and reliability were conducted.

Pregnancy-Specific Nausea and Vomiting Severity Scale (PUQE-24) consists of 3 questions:duration of nausea or stomach discomfort, number of vomiting episodes, and number of retching episodes. Answers to the questions are scored between 1 and 5 points. The total score of the scale is obtained by the sum of the scores of the answers given to the questions. The lowest possible score that can be obtained from the scale is 3 and the highest score is 15. If the total score obtained as a result of the PUQE-24 scoring system is 3-6, it is considered mild, 7-12 is considered moderate, and 13-15 is considered severe nausea and vomiting. The scale has no subdimensions. Cronbacha alpha value of the Turkish version of the scale is 0.75.

3.World Health Organization Quality of Life Scale: The WHOQOL-100 scale was developed with the participation of 15 centers from many countries. This scale allows cross-cultural comparisons. WHOQOL-100 was later abbreviated as WHOQOLBREF. WHOQOL-BREF consists of four sub-dimensions: physical domain, spiritual domain, social domain and environmental domain. The validity and reliability of the World Health Organization Quality of Life Scale 31 Short Form-Turkish Version (WHOQOL-BREF-TR) in Turkey was determined. WHOQOL-BREF-TR used in this study consists of 27 questions. For each question, there are options that can be scored between 1 and 5. The scale does not have a total score. The score range that can be obtained from each other sub-dimension is obtained by multiplying the arithmetic mean of that sub-dimension by 4. The score range that can be received for each sub-dimension is between 4-20. Increasing scores from the subscales indicate that the quality of life also increases

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 6-14 weeks of pregnancy
* Pregnant women between the ages of 20-40
* Pregnant women with complaints of nausea and vomiting
* Pregnant women who report their discomfort as 5 or above on the vas scale
* Pregnant women who have not been diagnosed with risky pregnancy
* Pregnant women who do not have any psychological disorders
* Pregnant women who voluntarily agreed to participate in the research

Exclusion Criteria:

* Coordination and language problems in the pregnant woman
* Wants to leave the study at any time
* Not wanting to participate in the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Enrollment: 74 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy-Unique Quantification of Emesis and Nausea (PUQE-24) | 3 months
  The degree of reduction in the severity of nausea and vomiting. The PUQE-24 (Pregnancy-Unique Quantification of Emesis and Nausea) scale is used, where each question is scored between 1 and 5. The total score is the sum of these three questions. Minimum Score: 3 (each question scoring 1) Maximum Score: 15 (each question scoring 5) These scores are used to rate the severity of nausea and vomiting in pregnancy. Lower scores indicate milder symptoms, while higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
WHOQOL-BREF (World Health Organization Quality of Life - BREF) | 3 months
  Evaluation of improvements in quality of life or psychological well-being, patient satisfaction with the treatment, and reduction in the need for pharmacological interventions. The WHOQOL-BREF (World Health Organization Quality of Life - BREF) scale is used, which comprises 26 items covering four domains: physical health, psychological health, social relationships, and environment. Each domain is scored between 0 and 100. Minimum Score: 0 (poorer quality of life) Maximum Score: 100 (better quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif Universty, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided